CLINICAL TRIAL: NCT02423161
Title: Prospective Intraoperative and Perioperative Ophthalmic Imaging With Optical Coherence Tomography: PIONEER Study
Brief Title: PIONEER: Intraoperative and Perioperative OCT Study
Acronym: PIONEER
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Justis Ehlers, Assistant Professor of Ophthalmology, The Cleveland Clinic
Other Study IDs: 11-787
Record Dates: First submitted 2015-04-08; First posted 2015-04-22 (Estimated); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Retinal Detachment; Epiretinal Membrane; Macular Hole; Fuchs Endothelial Dystrophy
Keywords: OCT; image-guided surgery; vitreoretinal surgery; corneal surgery
MeSH Terms: conditions — Retinal Detachment; Epiretinal Membrane; Retinal Perforations; Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
OCT provides high-resolution information regarding the anatomic structure of the tissues of the eye in a 2-dimensional and 3-dimensional view. Much of this information is not able to be recognized by a clinician. Utilizing this information during surgery will allow for ophthalmic surgeons to better understand how surgical procedures impact the anatomic structure of the eye.

DETAILED DESCRIPTION:
Over the last decade, optical coherence tomography (OCT) has become a critical component to the evaluation of ophthalmic disease. Similar to ultrasound, OCT uses light to reconstruct an image of the tissue of interest. In effect, OCT has become to function as a light biopsy, allowing clinicians to visualize subtle pathologic changes in the tissue, such as macular edema or subretinal fluid. The use of OCT in the clinic setting has become the standard for monitoring diseases such as macular degeneration and diabetic retinopathy. It has quickly become the most frequent ordered diagnostic test in ophthalmology.

Due to restraints in the size and structure of the imaging equipment, the use of OCT in the operating room has been limited. More recently, modifications to OCT table-top models as well as the development of hand-held OCT probes have allowed for the translation of OCT technology into the operating room. The high resolution anatomic information that is gained from OCT imaging is a natural complement to the ophthalmic surgeon. Using OCT during vitreoretinal surgery has revealed subtle changes in the microarchitecture of the retina in diseases such as retinal detachment, macular hole, and optic pit, that were not previously known. Using OCT during lamellar corneal transplant procedures, anterior segment surgeons have been able to image proper placement of the graft that was previously unattainable with a standard surgical microscopic view.

Using information gained from OCT, surgeons may be able to improve surgical decision making and improve clinical outcomes. For this study, subjects undergoing ophthalmic surgery, including vitreoretinal surgery and anterior segment surgery, would have OCT imaging performed in the perioperative period, intraoperative period, or both to document architectural changes in the ocular tissues. This information would be prospectively collected and reviewed for associations with anatomic and functional outcomes.

A microscope-mounted OCT system will be used to assess feasibility and utility of imaging during ophthalmic surgical milestones.

ELIGIBILITY:
Inclusion Criteria:

* The study population includes any patient requiring ophthalmic surgery

Exclusion Criteria:

* Children under the age of 18
* Cognitive/Mentally impaired or unable to provide consent
* Media opacity precluding OCT scanning

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes any patient requiring ophthalmic surgery
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2011-08; Primary Completion 2014-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Feasibility of intraoperative OCT | 3 years
  Defined as percentage of cases where OCT was successfully able to be obtained during surgery

SECONDARY OUTCOMES:
Utility of intraoperative OCT | 3 years
  Defined as percentage of cases where the OCT altered surgical decision-making based on surgeon-report on questionnaire
Safety of intraoperative OCT | 3 years
  Defined as the percentage of subjects that experience adverse events that were related to the intraoperative OCT and/or in excess of what might be expected relative to the surgery performed
Time requirements for intraoperative OCT | 3 years
  Defined as the mean number of minutes required to completed intraoperative imaging during a surgical case

CONTACTS AND LOCATIONS:
Overall Officials: Justis P Ehlers, MD, Principal Investigator — Cole Eye Institute, Cleveland Clinic, OH 44195
Locations (1):
- Cole Eye Institute, Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Background] Ehlers JP, Ohr MP, Kaiser PK, Srivastava SK. Novel microarchitectural dynamics in rhegmatogenous retinal detachments identified with intraoperative optical coherence tomography. Retina. 2013 Jul-Aug;33(7):1428-34. doi: 10.1097/IAE.0b013e31828396b7. PMID 23609120
- [Background] Ehlers JP, Xu D, Kaiser PK, Singh RP, Srivastava SK. Intrasurgical dynamics of macular hole surgery: an assessment of surgery-induced ultrastructural alterations with intraoperative optical coherence tomography. Retina. 2014 Feb;34(2):213-21. doi: 10.1097/IAE.0b013e318297daf3. PMID 23860560
- [Result] Ehlers JP, Itoh Y, Xu LT, Kaiser PK, Singh RP, Srivastava SK. Factors associated with persistent subfoveal fluid and complete macular hole closure in the PIONEER study. Invest Ophthalmol Vis Sci. 2014 Dec 18;56(2):1141-6. doi: 10.1167/iovs.14-15765. PMID 25525173
- [Result] Ehlers JP, Dupps WJ, Kaiser PK, Goshe J, Singh RP, Petkovsek D, Srivastava SK. The Prospective Intraoperative and Perioperative Ophthalmic ImagiNg with Optical CoherEncE TomogRaphy (PIONEER) Study: 2-year results. Am J Ophthalmol. 2014 Nov;158(5):999-1007. doi: 10.1016/j.ajo.2014.07.034. Epub 2014 Jul 29. PMID 25077834
- [Result] Juthani VV, Goshe JM, Srivastava SK, Ehlers JP. Association between transient interface fluid on intraoperative OCT and textural interface opacity after DSAEK surgery in the PIONEER study. Cornea. 2014 Sep;33(9):887-92. doi: 10.1097/ICO.0000000000000209. PMID 25055146
- [Derived] Au J, Goshe J, Dupps WJ Jr, Srivastava SK, Ehlers JP. Intraoperative Optical Coherence Tomography for Enhanced Depth Visualization in Deep Anterior Lamellar Keratoplasty From the PIONEER Study. Cornea. 2015 Sep;34(9):1039-43. doi: 10.1097/ICO.0000000000000508. PMID 26114817